CLINICAL TRIAL: NCT04182867
Title: Measuring the Cardio-metabolic Response to Diet Quality Modification During Night Work: Shift-eat (Night) Pilot Study
Brief Title: Measuring the Cardio-metabolic Response to Diet Quality Modification During Night Work.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment difficulties within the time frame
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Drum2019RG
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-03

CONDITIONS: Shift Work
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UK dietary guideline diet (Experimental): A 4-day diet (food and beverage provision for 3 meals and 2 snacks) will be provided along with an eating plan (time of each meal / snack). The experimental diet will meet UK dietary guidelines for fiber, salt, sugar, saturated fat, fruit and vegetable intake. Energy (calorie) requirements for each participant will be calculated from age, sex and weight of the participant. The diet will be consumed across 3 consecutive night shifts.
  Interventions: Other: Dietary intervention
- Shift worker diet (Other): A 4-day diet (food and beverage provision for 3 meals and 2 snacks) will be provided along with an eating plan (time of each meal / snack). Typical 'shift diet' based on previous research investigating what UK night workers eat. The 'shift diet' will contain ~15% energy from added sugar, 15g fiber, 2.5 portions fruit/vegetable, no whole grains. Required energy intake (calories) for each day to maintain their current body weight. Energy (calorie) requirements for each participant will be calculated from age, sex and weight of the participant.The diet will be consumed across 3 consecutive night shifts.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Dietary modification (provision of diet).

SUMMARY:
The aim of this pilot study is to investigate the acute impact of diet quality modification during night work on 24-hr glucose variability (GV) and heart rate variability (HRV) in healthy free-living employees.

DETAILED DESCRIPTION:
An increasing body of data reports deterioration of cardio-metabolic health in shift workers. For example, large scale meta-analyses have reported shift workers to be at increased risk of developing type 2 diabetes and of experiencing a coronary event, compared to day working employees.

Shift work causes complex changes in physiology (desynchrony of circadian rhythms) and behaviors including activity, sleep and eating patterns. The importance of meal timing is becoming increasingly recognized in both chronobiology and nutrition fields, with emerging awareness of 'chrono-nutrition', the interaction between nutrition and circadian time.

Given the importance to the economy of a healthy aging workforce, and the increase in shift work prevalence, it is important to establish if diet modification can reduce the health disparities between shift and day working employees.

ELIGIBILITY:
Inclusion Criteria:

* Current night shift worker (defined as a period of work between 11pm and 6am) working regular blocks of 3 night shifts.
* Body mass index between 18.5 and 35 kg/m2.
* Weight stable (no weight change by more than 3 kg in the last 2 months).
* Not a regular smoker (1 or more cigarettes per day) and would be willing not to smoke for the duration of the study.
* Not pregnant or breastfeeding.
* Not diagnosed with heart attack, stroke, angina, thrombosis, liver or kidney diseases, diabetes, chronic gastrointestinal disorder or cancer.
* Not currently taking medication to stabilize blood glucose (e.g. acarbose, metformin or sulfonylureas).
* Not started new medication within the last 3 months likely to interfere with energy metabolism, appetite regulation and hormonal balance, including: anti-inflammatory drugs or steroids, antibiotics, androgens, phenytoin, erythromycin or thyroid hormones.
* Do not take medication for blood pressure e.g. diuretics, (beta-blockers, Ca-channel, ACE inhibitors, Angiotensin Receptor blockers)
* Do not have diagnosed hypertension (high blood pressure, systolic blood pressure that is higher than 180 mmHg and or diastolic blood pressure that is higher than 110 mmHg).
* Not diagnosed with arterial fibrillation or any other condition that affects heart rate (e.g. arrhythmia).
* No food intolerance, allergies, hypersensitivity or follow any dietary restrictions (e.g. gluten intolerance, coeliac, lactose intolerance, vegan or vegetarian) that will prevent the ability to follow the test diets.
* Do not have a history substance abuse, or current high alcohol intake (>28 units/week for males and >21 units/week for females).
* Able to understand the information sheet and willing to comply with study protocol and able to follow dietary instructions before and during the study.
* Ability to prepare basic meals from ingredients provided.
* No travel arrangements outside UK within the period of data collection.
* Not already participating in a clinical trial.
* Able to give informed written consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose variability (mean amplitude of glycaemic excursions) | 3 night shifts, an average of 72 hours
  24-hr blood glucose variability measured by continuous glucose monitor
Blood glucose variability (coefficient variation) | 3 night shifts, an average of 72 hours
  24-hr blood glucose variability measured by continuous glucose monitor
Blood glucose variability (time in range) | 3 night shifts, an average of 72 hours
  24-hr blood glucose variability measured by continuous glucose monitor
Heart rate variability | 3 night shifts, an average of 72 hours
  24-hr heart rate variability measured by heart rate monitor

SECONDARY OUTCOMES:
Acceptability of test diet | 3 night shifts, an average of 72 hours
  Likert scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Life Course Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No